CLINICAL TRIAL: NCT00744757
Title: A Phase II Multi-center Study of 5-AZA-2'-Deoxycytidine (Decitabine) Single Agent in Taiwanese Patients With Myelodysplastic Syndrome (MDS)
Brief Title: An Efficacy and Safety Study of Decitabine in Participants With Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014785; DACOGENMDS2001
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Myelodysplastic Syndrome
Keywords: 5-aza-2'-deoxycytidine; decitabine; dacogen; Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Decitabine (Experimental): Decitabine 20 milligram per square meter (mg per m^2) will be administered intravenous (into a vein) infusion (a fluid or a medicine delivered into a vein by way of a needle) over 1 hour, once daily for 5 consecutive days of a 28 days cycle up to 8 cycles or continued until disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — Decitabine 20 mg per m^2 will be administered intravenous infusion over 1 hour, once daily for 5 consecutive days of a 28 days cycle up to 8 cycles or continued until disease progression or unacceptable toxicity.
  Other Names: Dacogen; 5-aza-2'-deoxycytidine

SUMMARY:
The purpose of this study is to evaluate the response rate of decitabine in previously treated and untreated Taiwanese participants with Myelodysplastic Syndrome (MDS - a disease associated with decreased production of blood cells, blood cells are produced but do not mature normally).

DETAILED DESCRIPTION:
This is an open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving, "unblinded"), multi-center (when more than 1 hospital or medical school team work on a medical research study), single-arm study of decitabine. The study will consist of 5 phases: Pre-treatment phase (before 30 days of first dose), Treatment phase (consist of 8 cycles, each cycle of 28 days), End-of-treatment phase (consist of 30-42 days after the last dose of cycle 8, or at time of discontinuation), Extension phase (1 cycle of 4 weeks) and Post-study phase or follow-up phase (every 2 months until 1 year, lost to follow-up or death). Participants who achieve a complete remission (when a medical problem gets better or goes away at least for a while) will be treated for at least 2 more cycles after first documentation of complete response (CR), after which treatment can be discontinued. Decitabine in a dose of 20 milligram per square meter (mg per m^2) will be administered intravenously over 1 hour infusion, 1 hour, once daily for 5 consecutive days of a 28 days cycle up to 8 cycles or continued until disease progression or unacceptable toxicity. The primary objective is to evaluate the best response rate (complete response and partial response). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented pathological (bone marrow, no longer than 30 days before first dosing in study) evidence of Myelodysplastic syndromes (MDS) or of chronic myelomonocytic leukemia (CMML) by World health organisation classification
* Participants with international prognostic scoring system (IPSS) score equal to 0.5 or more (only for participants for whom IPSS is applicable)
* Participants with an Eastern oncology cooperative group (ECOG) performance status of 0-2
* Participants with adequate hepatic (liver) and renal (kidney) function as measured by pre-treatment laboratory criteria within 21 days of starting treatment with decitabine
* Participants must have recovered from toxic effects of previous therapy and not receiving any chemotherapy for a minimum of 4 weeks (6 weeks if the participants has been treated with a nitrosoureas) before to the first dose of study drug

Exclusion Criteria:

* Participants with a diagnosis of acute myeloid leukemia (AML) (greater than 30 percent bone marrow blasts)
* Participants with AML with multilineage dysplasia (abnormal development or cell growth) following MDS (20-30 percent bone marrow blasts) can be enrolled. For these latter participants an observation period of 1 month is necessary to exclude those participants with rapid progression to full blown AML
* Participants with previous treatment with azacitadine or decitabine or hematopoietic stem cell transplantation less than 1 year prior to study enrollment
* Participants with past history of malignancy and received any treatment for this before malignancy within the last 3 years, except for superficial bladder cancer, basal cell or squamous cell carcinoma of the skin, cervical intraepithelial neoplasia (CIN) or prostate intraepithelial neoplasia (PIN)
* Participants with known hepatitis B (surface antigen-positive) or active hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-08; Primary Completion 2010-09 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd
Locations (6):
- Taiwan (6):
  - Changhua
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Tau-Yuan County 333

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Decitabine
Started | 37
Completed | 16
Not Completed | 21
Not completed — Objective disease progression | 7
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 1
Not completed — Death | 6
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine
Number analyzed (Participants) | 37
Age Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response
Description: Percentage of participants with response: complete response (CR) or partial response (PR) according to International Working Group (IWG) 2006 criteria was evaluated. CR in bone marrow is defined as<=to 5% myeloblasts with normal maturation of all cell lines and persistent dysplasia was noted in peripheral blood hemoglobin >=11 gram (g) per deciliter (dl), platelets >=100*10^9 liter (l), neutrophils >=1.0*10^9 l, Blasts 0%. Partial response is defined as all CR criteria if abnormal before treatment except: bone marrow blasts decreased by >=50% over pre-treatment but still >=5%.
Time Frame: Day 1 of Cycle 2, 4, 6, 8; each Cycle of 28 days and End of treatment (30-42 days after Cycle 8 or early withdrawal)
Population: The efficacy-evaluable (EE) population included all participants who received at least 2 cycles of treatment. Participants who died before receiving 2 complete cycles or were taken off study due to progressive disease were included. Here 'N' specifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Decitabine
Number analyzed (Participants) | 34
Percentage of Participants | 23.5

2. Secondary Outcome: Percentage of Participants With Hematologic Treatment Response
Description: Hematologic treatment response was assessed as per IWG 2006 criteria. This is measured in erythroid(HI-E), platelet(HI-P) and neutrophil(HI-N) lineages. HI-E response(pre-treatment<11 gram per deciliter [g/dl]):hemoglobin increase by>=1.5 g/dl and relevant reduction in RBC transfusions by 4 RBC transfusions/8week. HI-P response (pre-treatment<100*109/l):absolute increase of >=30*10^9/l for participants starting with>20*10^9/l and increase from <20*10^9/l to>20*10^9/l and by at least 100%. HI-N response (pre-treatment<1.0*10^9/l): at least 100% increase and an absolute increase >0.5*10^9/l.
Time Frame: Day 1 of Cycle 1, 2, 3, 4, 5, 6, 7 and 8, each Cycle of 28 days and End of treatment (30-42 days after Cycle 8 or early withdrawal)
Population: Intent-to-treat (ITT) population was defined as all participants who had received at least one dose of treatment. Here 'N' specifies those participants who were evaluable for this outcome measure and 'n' specifies those participants who were evaluable for this outcome measure at given time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Decitabine
Number analyzed (Participants) | 34
Percentage of participants
  Cycle 1: HI-E | 5.9
  Cycle 1: HI-P | 8.8
  Cycle 1: HI-N | 2.9
  Cycle 2: HI-E | 17.2
  Cycle 2: HI-P | 27.6
  Cycle 2: HI-N | 6.9
  Cycle 3: HI-E | 28.6
  Cycle 3: HI-P | 39.3
  Cycle 3: HI-N | 17.9
  Cycle 4: HI-E | 37.0
  Cycle 4: HI-P | 33.3
  Cycle 4: HI-N | 7.4
  Cycle 5: HI-E | 40.9
  Cycle 5: HI-P | 40.9
  Cycle 5: HI-N | 13.6
  Cycle 6: HI-E | 52.4
  Cycle 6: HI-P | 61.9
  Cycle 6: HI-N | 19.1
  Cycle 7: HI-E | 47.1
  Cycle 7: HI-P | 52.9
  Cycle 7: HI-N | 5.9
  Cycle 8: HI-E | 43.8
  Cycle 8: HI-P | 56.3
  Cycle 8: HI-N | 12.5
  End of treatment: HI-E | 27.6
  End of treatment: HI-P | 34.5
  End of treatment: HI-N | 6.9

3. Secondary Outcome: Percentage of Participants With Cytogenetic Response
Description: Cytogenetic responses was assessed as per IWG 2006 criteria which define complete response as disappearance of the chromosomal abnormality without appearance of new ones and partial response as at least 50 percent reduction of the chromosomal abnormality.
Time Frame: Day 1 of Cycle 2, 4, 6, 8; each Cycle of 28 days and End of treatment (30-42 days after Cycle 8 or early withdrawal)
Population: ITT population was defined as all participants who had received at least one dose of treatment. Here 'N' specifies those participants who were evaluated for this outcome measure and 'n' specifies those participants who were evaluated at given time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Decitabine
Number analyzed (Participants) | 20
Percentage of participants
  Cycle 2, Complete Response (n=18) | 22.2
  Cycle 2, Partial Response (n=18) | 0.0
  Cycle 4, Complete Response (n=20) | 20.0
  Cycle 4, Partial Response (n=20) | 25.0
  Cycle 6, Complete Response (n=11) | 18.2
  Cycle 6, Partial Response (n=11) | 27.3
  Cycle 8, Complete Response (n=6) | 0.0
  Cycle 8, Partial Response (n=6) | 0.0
  End of treatment, Complete Response (n=17) | 11.8
  End of treatment, Partial Response (n=17) | 5.9

4. Secondary Outcome: Time to Acute Myeloid Leukemia (AML) Progression or Death
Description: Time to AML is defined as greater than 30 percent of blasts in bone marrow or the time to death was calculated from the date of treatment start until disease progression to AML or until death, which ever occurred first. Participants who were still alive and did not progress to AML were censored at the moment of last visit.
Time Frame: Start of treatment until disease progression or death (whichever occur first) or up to 736 days
Population: ITT population was defined as all participants who had received at least 1 dose of study medication.
Measure: Median (Full Range); unit: Months
Arm/Group | Decitabine
Number analyzed (Participants) | 37
Months | 22.8 [0.3 to 25.4]

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of treatment start until death (whatever the cause). It was calculated from Kaplan-Meier estimates. Participants still alive were censored at the moment of last visit or contact.
Time Frame: Start of treatment until disease progression or death (whichever occur first) or up to 736 days
Population: ITT population was defined as all participants who had received at least 1 dose of study medication.
Measure: Median (Full Range); unit: Months
Arm/Group | Decitabine
Number analyzed (Participants) | 37
Months | 22.8 [0.3 to 25.4]

6. Secondary Outcome: Percentage of Participants With Transfusion Dependency
Description: Transfusion requirements for both red blood cells as well as platelets were recorded for each participant.
Time Frame: 8 weeks before first dose until disease progression or death (whichever occur first) or up to 736 days
Population: ITT population was defined as all participants who had received at least 1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Decitabine
Number analyzed (Participants) | 37
Percentage of participants | 100

7. Secondary Outcome: Percentage of Participants With Transfusion Independency
Description: Transfusion independent participants were calculated from all the participants who required transfusion in the duration of 8 weeks before first dose until disease progression or death or up to 736 days. Transfusion independence was defined as lack of requirement for transfusions for at least 8 weeks.
Time Frame: 8 weeks before first dose and 736 days of treatment
Population: ITT population was defined as all participants who had received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Decitabine
Number analyzed (Participants) | 37
percentage of participants | 27

8. Secondary Outcome: Duration for Hospitalization
Description: Duration of hospitalization was calculated for each participant, using the sum of all hospital days by subtracting the date of discharge from the date of admission.
Time Frame: Cycle 1 up to Cycle 8, each cycle of 28 days.
Population: ITT population was defined as all participants who had received at least one dose of treatment. Here 'n' specifies those participants who were evaluated for this outcome measure at given time point.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Decitabine
Number analyzed (Participants) | 37
Days
  Cycle 1 (n=37) | 9.0 (9.4)
  Cycle 2 (n=30) | 15.4 (16.2)
  Cycle 3 (n=28) | 13.3 (11.5)
  Cycle 4 (n=28) | 27.1 (52.9)
  Cycle 5 (n=22) | 22.5 (38.6)
  Cycle 6 (n=21) | 7.5 (5.0)
  Cycle 7 (n=17) | 33.3 (56.5)
  Cycle 8 (n=16) | 5.0 (0.0)

9. Secondary Outcome: Number of Events Which Led to Hospitalization
Description: The events (reasons) for hospitalizations such as infection, transfusion, acute choleycystitis, allergic transfusion reaction, dyspnoea with right pleural effusion, febrile neutropenia, fever, for decitabine, Myelodysplastic Syndrome (MDS) hematuria, paronychia, pneumonia, heart failure, peri-anal abscess (PAA), pancytopenia,fluctuated neutropenia fever, right dorsal foot cellulitis, Right lower (Rt.Lw) lung pneumonia with impending respiratory (resp) failure, Serious adverse event (SAE)+schedule hospitalization for decitabine, septic shock and not available were reported.
Time Frame: Start of treatment until disease progression or death or up to Cycle 8, each cycle of 28 days
Population: ITT population was defined as all participants who had received at least 1 dose of study medication.
Measure: Number; unit: Events
Arm/Group | Decitabine
Number analyzed (Participants) | 37
Events
  Infection | 10
  Transfusion | 4
  Acute choleycystitis | 1
  Allergic transfusion reaction | 1
  Dyspnoea with right pleural effusion | 4
  Febrile neutropenia | 16
  Fever | 4
  For Decitabine | 33
  MDS hematuria | 2
  Paronychia, pneumonia, heart failure | 1
  PAA,pancytopenia,fluctuated neutropenia fever | 1
  Right dorsal foot cellulitis | 1
  Rt Lw lung pneumonia with impending resp. failure | 1
  SAE+Schedule hospitalization for Decitabine | 4
  Septic shock | 1
  Not available | 36

10. Secondary Outcome: Quality of Life Assessment
Description: The quality of life was assessed by the questionnaire QLQ C-30 designed by European Organization for the Research and Treatment of Cancer (EORTC). EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer participants. Most questions used 4-point scale (1=Not at All' to 4=Very Much') and 2 questions: Q29 on overall health and Q30 on overall quality of life uses 7-point scale ranging from 1=Very Poor to 7=Excellent. Higher score indicates better quality of life.
Time Frame: Day 1 of Cycle 1 and Cycle 8 (each cycle of 28 days)
Population: ITT population was defined as all participants who had received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Decitabine
Number analyzed (Participants) | 37
Unit on a scale
  Baseline, Q29 | 4.4 (1.5)
  Baseline, Q30 | 4.9 (1.3)
  End of treatment, Q29 | 4.3 (1.7)
  End of treatment, Q30 | 4.5 (1.8)

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last medication
Arm/Group | Decitabine
Serious Adverse Events (participants affected / at risk) | 28/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine (N=37)
Febrile neutropenia (Blood and lymphatic system disorders) | 19
Anaemia (Blood and lymphatic system disorders) | 3
Pancytopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Bone marrow failure (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiac valve vegetation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 5
Multi-organ failure (General disorders) | 3
Induration (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatitis acute (Hepatobiliary disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 7
Septic shock (Infections and infestations) | 4
Anal abscess (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Pneumonia fungal (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 1
Escherichia bacterial (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Fungaemia (Infections and infestations) | 1
Hepatic infection (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pneumonia klebsiella (Infections and infestations) | 1
Splenic abscess (Infections and infestations) | 1
Splenic infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine (N=37)
Leucopenia (Blood and lymphatic system disorders) | 28
Anaemia (Blood and lymphatic system disorders) | 23
Neutropenia (Blood and lymphatic system disorders) | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 20
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 7
White blood cell disorder (Blood and lymphatic system disorders) | 5
Pancytopenia (Blood and lymphatic system disorders) | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Platelet disorder (Blood and lymphatic system disorders) | 3
Lymphadenitis (Blood and lymphatic system disorders) | 2
Splenomegaly (Blood and lymphatic system disorders) | 2
Cardiomegaly (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 3
Bradycardia (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Conjunctival haemorrhage (Eye disorders) | 4
Conjunctivitis (Eye disorders) | 3
Nausea (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 12
Mouth ulceration (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 10
Abdominal distension (Gastrointestinal disorders) | 8
Gingival bleeding (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 6
Haemorrhoids (Gastrointestinal disorders) | 6
Abdominal pain upper (Gastrointestinal disorders) | 5
Mouth haemorrhage (Gastrointestinal disorders) | 5
Melaena (Gastrointestinal disorders) | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Gingival pain (Gastrointestinal disorders) | 3
Haematochezia (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Dysgeusia (Gastrointestinal disorders) | 2
Reflux oesophagitis (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Gingivitis (Gastrointestinal disorders) | 2
Tongue haemorrhage (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 13
Fatigue (General disorders) | 13
Malaise (General disorders) | 13
Oedema peripheral (General disorders) | 13
Asthenia (General disorders) | 5
Chest discomfort (General disorders) | 4
Chest pain (General disorders) | 4
Oedema (General disorders) | 4
Chills (General disorders) | 3
Pain (General disorders) | 3
Hyperhidrosis (General disorders) | 2
Ulcer (General disorders) | 2
Hepatic cyst (Hepatobiliary disorders) | 3
Jaundice (Hepatobiliary disorders) | 2
Hypersensitivity (Immune system disorders) | 2
Pneumonia (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 8
Cellulitis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 5
Herpes simplex (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 3
Oral Candidiasis (Infections and infestations) | 3
Paronychia (Infections and infestations) | 2
Sepsis (Infections and infestations) | 3
Tinea pedis (Infections and infestations) | 3
Onychomycosis (Infections and infestations) | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 7
Wound complication (Injury, poisoning and procedural complications) | 4
Contusion (Injury, poisoning and procedural complications) | 3
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 2
Weight decreased (Investigations) | 6
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 4
Haemoglobin (Investigations) | 4
Monocyte count decreased (Investigations) | 3
Basophil count increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Cardiac murmur (Investigations) | 2
Eosinophil count increased (Investigations) | 2
Lymphocyte count increased (Investigations) | 2
Neutrophil count (Investigations) | 2
Urine output decrease (Investigations) | 2
Weight increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 14
Hypokalaemia (Metabolism and nutrition disorders) | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 5
Hyperbilirubinaemia (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 14
Headache (Nervous system disorders) | 7
Hypoaesthesia (Nervous system disorders) | 3
Poor quality sleep (Nervous system disorders) | 2
Vertigo (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 8
Anxiety (Psychiatric disorders) | 5
Depressed mood (Psychiatric disorders) | 3
Renal failure acute (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Acute tonsillitis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 11
Ecchymosis (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 6
Erythema (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Petechiae (Vascular disorders) | 5
Haematoma (Vascular disorders) | 3
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Periodontitis (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less